CLINICAL TRIAL: NCT04536545
Title: Evaluation of New Semen Collection & Transportation Kit in Maintaining the Quality of Semen Subjected to Overnight Shipping
Brief Title: Evaluation of New Semen Collection & Transportation Kit
Status: Completed | Type: Observational
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-729
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Sperm Parameters in Fertile and Infertile Men

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Examine the effect of overnight transport conditions on sperm parameters on semen samples collected and mailed to Cleveland Clinic Andrology center.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy men with normozoospermic semen parameters
* Infertile men referred by the infertility specialist (urologist)

Exclusion Criteria:

* Controls with abnormal semen parameters
* Infertile men from other referrals (Gynecologists)
* Severe oligozoospermic (<1 x 106 sperm/mL) infertile men

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Fertile and infertile men in the Cleveland area
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Sperm concentration | 24 hours
  Change in sperm concentration from 0 to 24 hours in millions per mL
Sperm motility | 24 hours
  Change in sperm motility from 0 to 24 hours in %
Sperm forward motility | 24 hours
  Change in sperm forward motility from 0 to 24 hours in %
Sperm morphology | 24 hours
  Change in sperm morphology from 0 to 24 hours using Kruger criteria

SECONDARY OUTCOMES:
Sperm concentration | 36 hours
  Change in sperm concentration from 0 to 36 hours in millions per mL
Sperm motility | 36 hours
  Change in sperm motility from 0 to 36 hours in %
Sperm forward motility | 36 hours
  Change in sperm forward motility from 0 to 36 hours in %
Sperm morphology | 36 hours
  Change in sperm morphology from 0 to 36 hours using Kruger criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Agarwal, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States